CLINICAL TRIAL: NCT05977257
Title: VitaFlow® Transcatheter Aortic Valve Replacement System Pre-market Trial Long Term Follow Up （VITAL）
Acronym: VITAL
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: VITAL-2023-192R
Record Dates: First submitted 2023-07-10; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non Interventional long term safety follow up: Non Interventional long term safety follow up
  Interventions: Device: VitaFlow® Transcatheter Aortic Valve Replacement System

INTERVENTIONS:
Device: VitaFlow® Transcatheter Aortic Valve Replacement System — This study is an observational study, for who have joined the VitaFlow® Catheter Aortic Valve System pre-market trial

SUMMARY:
This study is an observational study to evaluate the long-term safety and effectiveness of the valve system.

DETAILED DESCRIPTION:
This study is an observational study, for who have joined the VitaFlow® Catheter Aortic Valve System pre-market trial (Protocol No. valve -2014-04) in 4 designated research institutions, and follow-up from 6 to 10 years after the procedure, To evaluate the long-term safety and effectiveness of the valve system.

ELIGIBILITY:
Inclusion Criteria:

* Must meet 1, 2, 3, 4 or 1, 5 to be selected:

  1. Patients who have participated in the VitaFlow® transcatheter aortic valve system pre-market trial in the 4 designated research institutions*;
  2. Be able to get in touch with the patient or his legal guardian/relative;
  3. Patients who can understand the purpose and nature of the follow-up of this study, and are willing to cooperate with the follow-up and provide follow-up information;
  4. Sign the informed consent form;
  5. Patients who are known to have died.

     * 4 research institutions: Zhongshan Hospital Fudan University, Second Affiliated Hospital of Zhejiang University School of Medicine, West China Hospital of Sichuan University and Fuwai Hospital.

Exclusion Criteria:

1. Participate in clinical trials of other drugs or medical devices and have not yet reached the primary endpoint;
2. The investigator judges that the patient's compliance is poor and the study cannot be completed as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have participated in the VitaFlow® transcatheter aortic valve system pre-market trial
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 7years after the operation
  rate of all cause mortality

SECONDARY OUTCOMES:
Cardiac death | 6 years, 7 years, 8 years, 9 years and 10 years after the operation
  rate of Cardiac death
Stroke | 6 years, 7 years, 8 years, 9 years and 10 years after the operation
  rate of stroke
valve-related rehospitalization | 6 years, 7 years, 8 years, 9 years and 10 years after the operation
  rate of valve-related rehospitalization
Serious Adverse Event | 6 years, 7 years, 8 years, 9 years and 10 years after the operation
  rate of Serious Adverse Event
Blood pressure | 6 years, 7 years, 8 years, 9 years and 10 years after the operation
  Systolic and Diastolic Blood Pressure
The 12-Item Short Form Health Survey (SF-12) | 6years, 7years, 8 years, 9 years and 10 years after the operation
  Scores range from 0 to 100, higher scores are better
Mean transvalvular pressure gradient | 7years,and 10 years after the operation
  Transthoracic Echocardiogram test
Effective orifice area | 7years,and 10 years after the operation
  Transthoracic Echocardiogram test
Peak velocity | 7years,and 10 years after the operation
  Transthoracic Echocardiogram test
class of Paravalvular leak | 7years,and 10 years after the operation
  Transthoracic Echocardiogram test
class of Aortic regurgitation | 7years,and 10 years after the operation
  Transthoracic Echocardiogram test
New York Heart Association Class for heart function | 7years,and 10 years after the operation
  NYHA class
Kansas City Cardiomyopathy Questionnaire | 7years,and 10 years after the operation
  Kansas City Cardiomyopathy Questionnaire(score 0-100), higher scores are better
Natriuretic peptide tests ( NT Pro-BNP or BNP) | 7years,and 10 years after the operation
  blood test
moderate and severe structural valve deterioration SVD | 7years,and 10 years after the operation
  Transthoracic Echocardiogram test
bioprosthetic valve failure，BVF | 7years,and 10 years after the operation
  Transthoracic Echocardiogram test
All cause mortality | 6 years, 8 years, 9 years and 10 years after the operation
  rate of all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Daxin Zhou, Principal Investigator — Fudan University
Locations (4):
- China (4):
  - Fuwai CVD Hospital of Chinese Academy of Medical Sciences, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhongshan Hospital Fudan University, Shanghai